CLINICAL TRIAL: NCT00516932
Title: Pharmacogenomics of Antidepressant Response in Children and Adolescents
Acronym: PARCA
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00001300; P30MH066386-01 (NIH); DSIR CTM 4398; Pro00001300
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Anxiety Disorders; Depression; Eating Disorders; Obsessive-Compulsive Disorder; Suicide Prevention
Keywords: Suicidal Event; Behavioral Activation
MeSH Terms: conditions — Anxiety Disorders; Depression; Feeding and Eating Disorders; Obsessive-Compulsive Disorder; Suicide Prevention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary DNA retained at the Duke Center for Human Genetics
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will identify variations in genes that may be involved in the development of suicidal events or certain behaviors in youth who are exposed to antidepressant medications.

DETAILED DESCRIPTION:
Pharmacogenomics of Antidepressant Response in Children and Adolescents (PARCA) is a sub-study of the Antidepressant Safety in Kids (ASK) study. PARCA and ASK are part of the Child and Adolescent Psychiatry Trials Network (CAPTN).

Selective serotonin reuptake inhibitor (SSRI) and serotonin-norepinephrine reuptake inhibitor (SNRI) medications are prescribed to approximately 2 to 3% of American children. Evidence suggests that these medications are beneficial for treating obsessive-compulsive disorder (OCD), anxiety disorders, and major depressive disorder. Following hearings in February and September of 2004, the FDA mandated Black Box warnings for all antidepressants, cautioning prescribers about the risk of treatment-emergent suicidal tendency in children and adolescents treated with these drugs. Although prescribing waned somewhat following the warning, many children continue to receive SSRIs and SNRIs for a variety of conditions that do not have empirically validated alternative treatments. Therefore, there is a pressing need to clearly understand the safety, tolerability, and effectiveness of SSRIs and SNRIs in children and adolescents. This study will identify variations in differentially expressed genes that may be involved in the development of suicidal events and certain behaviors in youth exposed to antidepressant medications.

Specific aims of the study include the following:

1. To establish a genetic susceptibility database by creating a DNA repository of 120 patients with a prospectively identified "Suicidal Event" and 360 closely matched antidepressant-tolerant controls, including rigorous phenotypic characterization of these patients;
2. To establish a genetic susceptibility database by creating a DNA repository of 120 patients with prospectively identified "Behavioral Activation" and 360 closely matched antidepressant-tolerant controls, including rigorous phenotypic characterization of these patients;
3. To establish a genetic susceptibility database by creating a DNA repository of 120 patients with prospectively identified co-occurring "Suicidal Event and Behavioral Activation" and 360 closely matched antidepressant-tolerant controls, including rigorous phenotypic characterization of these patients;
4. To identify genetic polymorphisms responsible for the development of "Suicidal Events" using a candidate gene approach, including biosynthetic pathways, metabolizing enzymes, transporters, ion channels, and receptors;
5. To identify genetic polymorphisms responsible for the development of "Behavioral Activation" using a candidate gene approach, including biosynthetic pathways, metabolizing enzymes, transporters, ion channels, and receptors;
6. To use these data along with data from the parent study, ASK, to better understand the relationship between "Suicidal Events" and "Behavioral Activation."

Participants will include participants of the ASK study who want to participate in the PARCA study. Participants will use a self-collection kit to provide a saliva sample. The saliva sample will be mailed to the study center for DNA analysis. There will be no study visits.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Receiving treatment in an outpatient, residential, or in-patient setting
* Meets DSM-IV diagnostic criteria for at least one of the following disorders: anxiety disorder, depressive disorder, eating disorder, or obsessive-compulsive disorder
* Receiving a new prescription for an SSRI or SNRI to treat one of the above disorders
* A confirmed diagnosis of a "Suicidal Event" or "Behavioral Activation" or both following SSRI or SNRI exposure of at least 3 days duration
* Willing to provide a sample of saliva for DNA analysis
* English- or Spanish-speaking

Exclusion Criteria for Patients:

* Inpatient status IF the enrolling inpatient clinician will not continue to follow the patient for the duration of the study
* Sibling that is already enrolled in the study
* Imminently suicidal and unable to comply with a no-suicide contract or, in the opinion of the treating clinician, has inadequate family monitoring for suicidality
* Acutely psychotic at study entry
* A demonstrated lack of benefit from or intolerance to SSRI/SNRI antidepressants, as a class
* Receiving treatment with a tricyclic antidepressant (TCA) at study enrollment, with the exception of low doses for enuresis for chronic pain. Patients may receive adjunctive TCA treatment during the study at the clinician's discretion.
* Received a monoamine oxidase inhibitor (MAOI), such as isocarboxazid (Marplan), phenelzine (Nardil), or tranylcypromine (Parnate), within the past 30 days
* Parasuicidal behavior or milder forms of suicidality or activation that do not meet the diagnostic criteria
* Refusal to participate in the pharmacogenomic study
* For bipolar depressed patients, a mixed- or manic-state at study entry without stable treatment with a mood stabilizer for manic symptoms
* Patient or family is unable to comply with the protocol

Note: Tolerant controls will be ineligible if they have a past history of a treatment-emergent "Suicidal Event" or "Behavioral Activation"

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Males and Females
  Age 7 -17 years
  Pre-specified disorder of anxiety disorder, depressive disorder, eating disorder, or obsessive-compulsive disorder.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Suicidal Event(120 patients) Behavioral Activation(120 patients) Co-occurring Suicidal Event + Behavioral Activation (120 patients) Tolerant controls (at a control to case ratio of 3:1) no evidence of Suicidal Events or Behavioral Activation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: John S. March, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Child and Adolescent Psychiatry Trials Network (CAPTN), Durham, North Carolina, United States

REFERENCES:
- See also: Click here for the ASK study, a related trial within the CAPTN network — http://www.clinicaltrials.gov/ct/show/NCT00395213